CLINICAL TRIAL: NCT03566797
Title: Secondary Sclerosing Cholangitis in Critically Ill Patients (SC-CIP): A Prospective Cohort Study
Brief Title: Secondary Sclerosis Cholangitis Prospective
Acronym: SSCpro
Status: Recruiting | Type: Observational
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Other Study IDs: SC_prospective
Record Dates: First submitted 2018-05-07; First posted 2018-06-25 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Secondary Sclerosis Cholangitis in Critically Ill Patients

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA, serum, plasma, stool urine
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- SC-CIP: Patients developing SC-CIP
- noSC-CIP: Patients with similar severity of critical illness not developing SC-CIP

SUMMARY:
SC-CIP is increasing in patients after critical illness. Pathogenesis is still largely unclear. Gut microbiome composition, gut permeability, bacterial translocation, inflammation and/or genetic variants contribute to the pathogenesis The aim of this project is to study gut microbiome composition, gut permeability, bacterial translocation, inflammation, bile acid composition and genetic polymorphisms by conducting a prospective cohort study in patients with a high risk to develop SC-CIP.

DETAILED DESCRIPTION:
Secondary sclerosing cholangitis in critically ill patients (SC-CIP) is a rare, quickly progressive, cholestatic liver disease which is observed in patients suffering from a severe illness with the need for long term treatment on an intensive care unit (ICU). Invasive ventilation, polytrauma, hypotension, systemic inflammatory response syndrome, burns, complex operations and severe (co-) morbidities such as obesity have been discussed as risk factors. Patients suffering from SC-CIP do not have any underlying liver disease. Usually, long- term ICU treatment is described as the trigger mechanism for the development of this disease, although also rapid development of SC-CIP after an ICU stay as short as nine days is described in a single case.

The pathogenesis of SC-CIP is not fully understood yet: Ischemic injury of the intrahepatic biliary system, bile cast formation and recurrent biliary infections are discussed as major factors. The disease leads to a progressive destruction of the intra- and extrahepatic biliary tree with the development of strictures resulting in liver fibrosis with in some cases rapid progression to cirrhosis with the need for liver transplantation within months. The gold standard for diagnosis is endoscopic retrograde cholangiopancreaticography (ERCP), although magnetic resonance cholangiopancreatography (MRCP) as non-invasive alternative can lead to the diagnosis in most cases. Prognosis is poor and transplant-free survival has been found to be 40 months in average. Liver transplantation is the only curative treatment, which shows excellent outcome and quality of life comparable to other indication for liver transplantation.

Microbiological analysis of bile from patients with SC-CIP and primary sclerosing cholangitis (PSC) show a significant different microbiological profile in these two cohorts with dominance of drug resistant organisms in the bile of SC-CIP. No data on the gut microbiome in SC-CIP are available so far. Other chronic liver diseases show distinct changes in microbiome composition with potential influence on the inflammation process in these liver diseases (non-alcoholic fatty liver disease (NAFLD), alcoholic liver disease, PSC and liver cirrhosis). In general a decrease in diversity, a higher abundance of potentially pathogenic species and a lower abundance of beneficial species has been observed.

Dysbiosis is thought to increase intestinal permeability. Increased gut permeability is most frequently observed in liver cirrhosis but was also found in alcohol-induced injury, NAFLD and hepatitis C-mediated liver injury. With an impaired gut permeability bacteria from the intestinal lumen can be translocated into extraintestinal parts of the body (lymph nodes, blood) and prompt inflammatory responses. Genetic polymorphisms in the Nucleotide-binding oligomerization domain-containing protein 2 (NOD2) gene, a known risk factor for bacterial translocation, increases the odds of developing SC-CIP.

It is hypothesized that the gut microbiome composition is altered in SC-CIP and that this is associated with increased gut permeability and markers of inflammation. Reasons for this might lie in gene polymorphisms influencing bacterial translocation or bile acid composition.

The aim of this study is to prospectively assess the incidence of SC-CIP in a cohort of patients at risk for developing SC-CIP (ICU treatment with the need for mechanical ventilation or extracorporeal membrane oxygenation >/= 5 days) and study differences in gut microbiome composition, gut permeability, bacterial translocation, inflammation as well as genetic polymorphisms in patients developing SC-CIP and patients with comparable disease severity who did not develop SC-CIP.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study OR "surrogate consent" by the institutional review board.
* Age above 18 years
* Mechanical ventilation or extracorporeal membrane oxygenation >/= 5 days

Exclusion Criteria:

* Primary or secondary sclerosing cholangitis diagnosed before current ICU admission

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to Intensive Care Units at the University Hospital Graz
Sampling Method: Probability Sample
Enrollment: 380 (Estimated)
Dates: Start 2018-07-20 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of SC-CIP in patients at risk | during hospital stay, on average 4 weeks
  risk is defined as need for mechanical ventilation or extracorporeal membrane oxygenation >/= 5 days

SECONDARY OUTCOMES:
Gut microbiome composition | at inclusion
  16S rRNA sequencing
Stool zonulin | at inclusion
  gut permeability marker, ELISA
Stool calprotectin | at inclusion
  gut inflammation marker, ELISA
Serum endotoxin | at inclusion
  bacterial translocation marker, cell-based assay
Serum lipopolysaccharide binding protein | at inclusion
  bacterial translocation marker, ELISA
soluble cluster of differentiation 14 (sCD14) | at inclusion
  bacterial translocation marker, ELISA
bile acid transporter polymorphisms | at inclusion
  sequencing of bile acid transporter genes
NOD2 polymorphisms | at inclusion
  sequencing of the NOD2 gene

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University Graz, Graz, Austria